CLINICAL TRIAL: NCT04636437
Title: Doravirine for Obese Persons on Integrase Inhibitors and Tenofovir Alafenamide (The Do IT Study)
Brief Title: Doravirine for Obese Persons on Integrase Inhibitors and Tenofovir Alafenamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5391; UM1AI068636 (NIH)
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — doravirine; emtricitabine tenofovir alafenamide; Racivir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DOR 100 mg + TAF/FTC (Experimental): By mouth daily with or without food
  Interventions: Drug: Doravirine 100 Mg; Drug: Integrase strand transfer inhibitors
- DOR 100 mg + TDF/FTC (Experimental): By mouth daily with or without food
  Interventions: Drug: Doravirine 100 Mg; Drug: tenofovir disproxil fumarate/emtricitabine
- Continuation of INSTI+TAF/FTC (Active Comparator): By mouth daily with or without food
  Interventions: Drug: Integrase strand transfer inhibitors; Drug: Tenofovir alafenamide/emtricitabine

INTERVENTIONS:
Drug: Doravirine 100 Mg — Participants received a 100 mg tablet by mouth daily with or without food.
  Other Names: DOR
  Arms: DOR 100 mg + TAF/FTC; DOR 100 mg + TDF/FTC
Drug: Integrase strand transfer inhibitors — INSTIs were acquired through the standard of care locally.
  Other Names: INSTI
  Arms: Continuation of INSTI+TAF/FTC; DOR 100 mg + TAF/FTC
Drug: Tenofovir alafenamide/emtricitabine — NRTIs (TAF/FTC) were acquired through the standard of care locally.
  Other Names: TAF, FTC
  Arms: Continuation of INSTI+TAF/FTC
Drug: tenofovir disproxil fumarate/emtricitabine — NRTIs (TDF/FTC) were acquired through the standard of care locally.
  Other Names: TDF, FTC
  Arms: DOR 100 mg + TDF/FTC

SUMMARY:
The purpose of this study was to determine if people with HIV and obesity taking an antiretroviral treatment regimen containing an integrase strand transfer inhibitor (INSTI) with (tenofovir alafenamide/emtricitabine (TAF/FTC) would either slow their rate of weight gain, or even lose weight, over the span of about 1 year after a switch to a regimen containing doravirine (DOR; a newer, non-nucleoside reverse transcriptase inhibitor medication) combined with either TAF/TFC or tenofovir disoproxil fumarate (TDF)/FTC.

DETAILED DESCRIPTION:
The study evaluated whether a switch from an INSTI to a DOR-based regimen would result in less weight gain or weight loss at 48 weeks among obese individuals with HIV and a suppressed viral load. The study also evaluated whether an additional switch from TAF/FTC to TDF/FTC, both in combination with DOR, had an effect on weight over 48 weeks. Participants enrolled in A5391 were taking INSTI-class medications, including bictegravir (BIC), dolutegravir (DTG), or raltegravir (RAL), all in combination with TAF/FTC. Additionally, the study examined whether a change in the HIV treatment regimen affects other health indicators, including waist circumference, metabolic and cardiovascular disease markers, body composition (fat and lean mass), bone density, and maintenance of virologic suppression. Finally, the study looked at the safety and tolerability of DOR with either TAF/FTC or TDF/FTC.

As originally designed, the trial's target population included individuals with an unintentional >10% weight gain in the 1-3 years after initiating or switching to an INSTI-based treatment regimen. Due to not meeting accrual targets during the first year of enrollment (July 2021 - July 2022), the trial protocol was updated to amend the target population (and associated eligibility criteria) to individuals with obesity (a screening body mass index [BMI] of ≥30 kg/m2) irrespective of weight history on INSTI-based ART. This update was implemented on November 17, 2022, at which time 64 participants had enrolled under the original trial design. The remaining participants enrolled using the revised eligibility criterion.

At a planned interim analysis in 2023, the method of blinded sample size re-estimation was used to assess if the trial's primary objective could be met with a sample size smaller than originally planned (n=222). Based on the pooled (e.g. over all arms) standard deviation of the primary outcome (weight change at 48 weeks), 150 participants would provide over 80% statistical power to detect the originally hypothesized 5% points change in weight between arms, assuming that this interim estimate was representative of the true variability about the primary outcome. As a result, the accrual goal was adjusted accordingly. The trial closed to enrollment in October 2024, having reached 147 participants.

ELIGIBILITY:
Inclusion Criteria:

Ability and willingness of participant or legal guardian/representative to provide informed consent.

HIV-1, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, or plasma HIV-1 RNA viral load. If a rapid HIV test or any FDA-approved HIV-1 E/CIA test kit is not available, two HIV-1 RNA values ≥2000 copies/mL at least 24 hours apart may be performed by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or by any non-US laboratory that is DAIDS Good Clinical Laboratory Practice (GCLP) compliant and, if performing HIV-1 RNA testing, is Virology Quality Assurance (VQA)-certified.

Currently on a bictegravir (BIC), dolutegravir (DTG), or raltegravir (RAL) + TAF/FTC regimen with ≥48 weeks prior to study entry.

Ability to acquire NRTIs (TAF/FTC or TDF/FTC) and INSTI through usual care for the duration of the study.

A BMI ≥30 kg/m2 at screening. No known plans to change or to initiate medications known to be associated with significant weight changes during study period.

Agree to adhere to assigned ART during the study period At least one HIV-1 RNA level <50 copies/mL (or below the lower limit of HIV-1 RNA detection available at the site if the lower limit of detection is >50) performed in the 48 weeks prior (≤48 weeks) to study screening, and at least one HIV-1 RNA level <50 copies/mL ≥48 weeks prior to study screening, using an FDA-approved assay performed by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that is VQA certified.

Screening HIV-1 RNA <50 copies/mL (or below the lower limit of HIV-1 RNA detection available if the lower limit of detection is >50) performed within 45 days prior to study entry by any US laboratory that possesses a CLIA certification or its equivalent, or at any network-approved non-US laboratory that is VQA certified.

For participants capable of becoming pregnant, negative serum or urine pregnancy test within 45 days prior to study entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or is using a point of care (POC)/ CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

Participants engaging in sexual activity and capable of becoming pregnant must agree to use contraception while on study drug (approximately 48 weeks) and for 8 weeks after the end of the study. At least one of the following contraceptive methods must be used:

* Intrauterine device (IUD)
* Hormone-based contraceptive
* Partner sterilization (i.e., vasectomy) and is the sole partner for the participant.

Transgender participants who are currently taking hormones must be on a stable hormone dose for >12 weeks prior to study entry. Transgender participants should not have active plans to change their hormone regimen or dose during the study period.

The following laboratory values obtained within 45 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate external quality assurance programs:

* Absolute neutrophil count (ANC) >750 cells/mm3
* Hemoglobin >10 g/dL for males and >9 g/dL for females (based on sex at birth)
* Calculated creatinine clearance ≥50 mL/min as estimated by the CKD-EPI equation (a calculator is available at: https://qxmd.com/calculate/calculator_251/egfr-using-ckd-epi)
* Aspartate aminotransferase (AST) (SGOT) <3x ULN
* Alanine aminotransferase (ALT) (SGPT) <3x ULN

Exclusion Criteria:

Historical or current evidence of the K65R/E/N or M184V/I mutations (for participants who have undergone HIV-1 genotyping), due to the potential for viral rebound after switch from an INSTI- to NNRTI-based regimen.

Historical or current evidence of major mutations associated with NNRTI resistance.

History of prior virologic failure in the opinion of the site investigator. For example, a confirmed plasma HIV-1 RNA >1000 copies/mL after having achieved viral suppression.

Prior exposure to single-dose nevirapine for the prevention of parent-to-child transmission of HIV.

Any history of significant renal toxicity while taking TDF (as determined by the site investigator).

Currently breast-feeding or pregnant, or intending to become pregnant during the duration of the study.

Current use, use in the 4 weeks preceding study entry, or anticipated use of prohibited drugs during the study period.

Anticipated start or cessation of any of the following drugs during the study period:

* Antipsychotics (e.g., clozapine, olanzapine, risperidone, etc.) and antidepressants (tricyclic antidepressants, e.g., amitriptyline, nortriptyline, etc.; selective serotonin reuptake inhibitors, e.g., fluoxetine, paroxetine, sertraline, etc.; and monoamine oxidase inhibitors, e.g., selegiline) associated with weight gain
* Anticonvulsants/mood stabilizers associated with weight gain (e.g., lithium, valproic acid) or weight loss (e.g., topiramate)
* Thyroid replacement hormones
* Anti-diabetic agents known to cause weight loss (e.g., GLP-1 receptor agonists such as exenatide, dulaglutide, semaglutide, metformin, and SGLT-2 inhibitors such as canagliflozin, dapagliflozin, etc.).

Planning to undergo bariatric surgery or initiate significant dietary or exercise changes within the study period (e.g., structured weight loss programs such as Weight Watchers), as determined by participant report.

Known allergy/sensitivity or any hypersensitivity to components of study drug or its formulation.

Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with ability to adhere to study requirements, or cessation of regular methamphetamine use, as determined by the site investigator, within 60 days prior to study entry.

Acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry.

A history of a diagnosis of osteoporosis or osteopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koethe, Study Chair — Vanderbilt University Medical Center
Locations (27):
- United States (27):
  - Alabama CRS (31788), Birmingham, Alabama
  - UCLA CARE Center CRS (601), Los Angeles, California
  - UCSD Antiviral Research Center CRS (701), San Diego, California
  - Ucsf Hiv/Aids Crs (801), San Francisco, California
  - Harbor-UCLA CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Whitman-Walker Institute, Inc. CRS (31791), Washington D.C., District of Columbia
  - The Ponce de Leon Center CRS (5802), Atlanta, Georgia
  - Northwestern University CRS (2701), Chicago, Illinois
  - Johns Hopkins University CRS (201), Baltimore, Maryland
  - Massachusetts General Hospital (MGH) CRS (101), Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS (107), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS (2101), St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS (31786), Newark, New Jersey
  - Weill Cornell Chelsea CRS (7804), New York, New York
  - Columbia Physicians and Surgeons (P&S) CRS (30329), New York, New York
  - Weill Cornell Upton CRS (7803), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Chapel Hill CRS (3201), Chapel Hill, North Carolina
  - Greensboro CRS (3203), Greensboro, North Carolina
  - Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Ohio State University CRS (2301), Columbus, Ohio
  - Penn Therapeutics CRS (6201), Philadelphia, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS (3652), Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington Positive Research CRS (1401), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the Advancing Clinical Therapeutics Globally (ACTG) by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the ACTG.
  * For what types of analyses? To achieve aims in the proposal approved by the ACTG.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the ACTG "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an ACTG Data Use Agreement before receiving the data."

REFERENCES:
- See also: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (Corrected Version 2.1 - July 2017) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (Version 2.0 - January 2010) — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: CKD-EPI Creatinine Equation (2021) — https://www.kidney.org/ckd-epi-creatinine-equation-2021-0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from July 27, 2021 to November 30, 2023 at 27 sites in the US.
Groups:
- DOR 100 mg + TAF/FTC: By mouth daily with or without food.
  Participants received a Doravirine 100 mg tablet by mouth daily.
  NRTIs (TAF/FTC) were acquired through the standard of care locally.
- DOR 100 mg + TDF/FTC: By mouth daily with or without food.
  Participants received a Doravirine 100 mg tablet by mouth daily.
  NRTIs (TDF/FTC) were acquired through the standard of care locally.
- Continuation of INSTI+TAF/FTC: By mouth daily with or without food.
  INSTIs and NRTIs (TAF/FTC) were acquired through the standard of care locally.
Period: Overall Study
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Started | 49 | 49 | 49
Completed | 39 | 45 | 43
Not Completed | 10 | 4 | 6
Not completed — Eligibility failure discovered after study entry | 2 | 1 | 0
Not completed — Started weight loss drug/program | 2 | 1 | 1
Not completed — Lost to Follow-up | 3 | 1 | 4
Not completed — Participant or physician decision | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was done in the treated population. This includes all participants who received at least one dose of their randomized study treatment. Two participants on the DOR 100mg + TAF/FTC arm did not start treatment and are not included.
Groups:
- DOR 100 mg + TAF/FTC: By mouth daily with or without food. Participants will receive a Doravirine 100 mg tablet by mouth daily. NRTIs (TAF/FTC) will be acquired through the standard of care locally.
- DOR 100 mg + TDF/FTC: By mouth daily with or without food. Participants will receive a Doravirine 100 mg tablet by mouth daily. NRTIs (TDF/FTC) will be acquired through the standard of care locally.
- Continuation of INSTI+TAF/FTC: By mouth daily with or without food. INSTIs and NRTIs (TAF/FTC) will be acquired through the standard of care locally.
- Total: Total of all reporting groups
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC | Total
Number analyzed (Participants) | 47 | 49 | 49 | 145
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [36 to 57] | 50 [39 to 55] | 52 [42 to 58] | 49 [40 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 24 | 71
  Male | 24 | 25 | 25 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 5 | 26
  Not Hispanic or Latino | 36 | 38 | 43 | 117
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 24 | 26 | 27 | 77
  White | 22 | 21 | 19 | 62
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 49 | 49 | 145
Weight [Median (Inter-Quartile Range); unit: kg] | 107.3 [90.4 to 124.8] | 95.9 [89.7 to 120.7] | 101.3 [92.7 to 113.0] | 99.7 [91.2 to 117.8]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 36.9 [33.2 to 41.3] | 34.4 [31.7 to 39.3] | 34.9 [32.3 to 39.2] | 34.9 [32.3 to 39.3]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Percent) in Body Weight (kg) From Entry to Week 48
Description: The percentage change is defined as weight at week 48 minus weight at entry, then divided by weight at entry, then multiplied by 100.
  Mean and confidence interval (CI) come from a linear regression model adjusting for entry weight, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: Analysis was done in the eligible treated population with data available at all timepoints. The eligible treated population includes all participants who received at least one dose of randomized study treatment and who were eligible as per eligibility criteria.
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 39 | 45 | 43
relative change % | -0.47 [-2.09 to 1.14] | -2.73 [-4.22 to -1.23] | -1.84 [-3.37 to -0.3]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in body weight from entry to week 48; Test type: Superiority; p = 0.23, Regression, Linear — Bonferroni adjustment for 2 pairwise comparisons of DOR-containing arms versus continuation of INSTI. Two sided 2.5% alpha; Mean Difference (Net) = 1.36, 97.5% CI 2-sided [-1.20 to 3.92] — Mean difference and CI come from a linear regression model adjusting for entry weight, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in body weight from entry to week 48; Test type: Superiority; p = 0.41, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.89, 97.5% CI 2-sided [-3.34 to 1.57] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change (Percent) in Body Weight (kg) From Entry to Week 24
Description: The percentage change is defined as weight at week 24 minus weight at entry, then divided by weight at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry weight, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 44 | 47 | 45
relative change % | 0.44 [-0.69 to 1.56] | -2.37 [-3.46 to -1.29] | -0.39 [-1.50 to 0.72]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in body weight from entry to week 24; Test type: Superiority; p = 0.31, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.83, 97.5% CI 2-sided [-0.99 to 2.64] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in body weight from entry to week 24; Test type: Superiority; p = 0.012, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.99, 97.5% CI 2-sided [-3.76 to -0.21] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change (Absolute) in Waist Circumference From Entry to Week 48
Description: The absolute change is defined as waist circumference at week 48 minus waist circumference at entry.
  Mean and CI come from a linear regression model adjusting for entry waist circumference, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 39 | 45 | 43
cm | 1.70 [-0.22 to 3.62] | -1.51 [-3.30 to 0.28] | -0.02 [-1.85 to 1.82]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in waist circumference from entry to week 48; Test type: Superiority; p = 0.20, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.72, 97.5% CI 2-sided [-1.33 to 4.77] — Mean difference and CI come from a linear regression model adjusting for entry waist circumference, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.25, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.49, 97.5% CI 2-sided [-4.43 to 1.44] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Mean Change (Absolute) in Waist Circumference From Entry to Week 24
Description: The absolute change is defined as waist circumference at week 24 minus waist circumference at entry.
  Mean and CI come from a linear regression model adjusting for entry waist circumference, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 43 | 47 | 45
cm | 1.03 [-0.88 to 2.94] | -0.29 [-2.11 to 1.54] | 1.19 [-0.68 to 3.06]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in waist circumference from entry to week 24; Test type: Superiority; p = 0.90, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.16, 97.5% CI 2-sided [-3.23 to 2.90] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.26, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.48, 97.5% CI 2-sided [-4.47 to 1.51] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Mean Change (Absolute) in Fasting Triglycerides From Entry to Week 48
Description: The absolute change is defined as triglycerides at week 48 minus triglycerides at entry.
  Mean and CI come from a linear regression model adjusting for entry triglycerides, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 37 | 43 | 43
mg/dL | 1.23 [-13.7 to 16.19] | -7.07 [-21.0 to 6.86] | 0.03 [-13.9 to 13.93]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting triglycerides from entry to week 48; Test type: Superiority; p = 0.91, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.19, 97.5% CI 2-sided [-22.2 to 24.59] — Mean difference and CI come from a linear regression model adjusting for entry fasting triglycerides, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.48, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -7.10, 97.5% CI 2-sided [-29.7 to 15.47] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Mean Change (Absolute) in Fasting Triglycerides From Entry to Week 24
Description: The absolute change is defined as triglycerides at week 24minus triglycerides at entry.
  Mean and CI come from a linear regression model adjusting for entry triglycerides, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 44 | 45 | 43
mg/dL | 2.21 [-18.3 to 22.69] | -1.10 [-21.4 to 19.17] | 17.42 [-3.31 to 38.16]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting triglycerides from entry to week 24; Test type: Superiority; p = 0.30, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.2, 97.5% CI 2-sided [-48.6 to 18.20] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.21, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -18.5, 97.5% CI 2-sided [-51.8 to 14.76] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Mean Change (Absolute) in Fasting Low-density Lipoprotein (LDL) Cholesterol From Entry to Week 48
Description: The absolute change is defined as LDL at week 48 minus LDL at entry. Mean and CI come from a linear regression model adjusting for entry LDL, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 37 | 43 | 42
mg/dL | -4.89 [-12.2 to 2.40] | -8.92 [-15.7 to -2.18] | -2.04 [-8.93 to 4.84]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting LDL from entry to week 48; Test type: Superiority; p = 0.58, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.84, 97.5% CI 2-sided [-14.4 to 8.72] — Mean difference and CI come from a linear regression model adjusting for entry fasting LDL, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting LDL from entry to week 48; Test type: Superiority; p = 0.16, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -6.88, 97.5% CI 2-sided [-18.0 to 4.20] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Mean Change (Absolute) in Fasting Low-density Lipoprotein (LDL) Cholesterol From Entry to Week 24
Description: The absolute change is defined as LDL at week 24 minus LDL at entry. Mean and CI come from a linear regression model adjusting for entry LDL, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 44 | 45 | 42
mg/dL | 0.24 [-5.31 to 5.79] | -11.9 [-17.4 to -6.40] | 3.16 [-2.57 to 8.89]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting LDL from entry to week 24; Test type: Superiority; p = 0.47, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -2.92, 97.5% CI 2-sided [-12.1 to 6.27] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting LDL from entry to week 24; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.1, 97.5% CI 2-sided [-24.2 to -5.91] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Mean Change (Absolute) in Fasting High-density Lipoprotein (HDL) Cholesterol From Entry to Week 48
Description: The absolute change is defined as HDL at week 48 minus HDL at entry. Mean and CI come from a linear regression model adjusting for entry HDL, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 37 | 43 | 43
mg/dL | 3.56 [-0.86 to 7.98] | -2.71 [-6.77 to 1.36] | 2.75 [-1.34 to 6.85]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting HDL from entry to week 48; Test type: Superiority; p = 0.79, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.80, 97.5% CI 2-sided [-6.17 to 7.77] — Mean difference and CI come from a linear regression model adjusting for entry fasting HDL, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting HDL from entry to week 48; Test type: Superiority; p = 0.063, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -5.46, 97.5% CI 2-sided [-12.1 to 1.16] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Mean Change (Absolute) in Fasting High-density Lipoprotein (HDL) Cholesterol From Entry to Week 24
Description: The absolute change is defined as HDL at week 24 minus HDL at entry. Mean and CI come from a linear regression model adjusting for entry HDL, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 44 | 45 | 43
mg/dL | -0.23 [-1.96 to 1.49] | -4.31 [-6.00 to -2.61] | 1.15 [-0.60 to 2.90]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting HDL from entry to week 24; Test type: Superiority; p = 0.27, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.38, 97.5% CI 2-sided [-4.21 to 1.45] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting HDL from entry to week 24; Test type: Superiority; p < 0.001, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -5.45, 97.5% CI 2-sided [-8.25 to -2.66] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Mean Change (Absolute) in Fasting Glucose From Entry to Week 48
Description: The absolute change is defined as glucose at week 48 minus glucose at entry. Mean and CI come from a linear regression model adjusting for entry glucose, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 37 | 43 | 42
mg/dL | 5.43 [-2.12 to 12.98] | -1.35 [-8.37 to 5.66] | 3.88 [-3.22 to 10.97]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting glucose from entry to week 48; Test type: Superiority; p = 0.77, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.55, 97.5% CI 2-sided [-10.3 to 13.44] — Mean difference and CI come from a linear regression model adjusting for entry fasting glucose, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.30, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -5.23, 97.5% CI 2-sided [-16.7 to 6.20] — [estimate comment as in outcome 11, analysis 1]

12. Secondary Outcome: Mean Change (Absolute) in Fasting Glucose From Entry to Week 24
Description: The absolute change is defined as glucose at week 24 minus glucose at entry. Mean and CI come from a linear regression model adjusting for entry glucose, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 43 | 45 | 43
mg/dL | 2.31 [-3.21 to 7.84] | -4.19 [-9.60 to 1.12] | 2.13 [-3.40 to 7.66]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting glucose from entry to week 24; Test type: Superiority; p = 0.96, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.18, 97.5% CI 2-sided [-8.78 to 9.15] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.11, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -6.32, 97.5% CI 2-sided [-15.2 to 2.55] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Mean Change (Absolute) in Fasting Insulin From Entry to Week 48
Description: The absolute change is defined as insulin at week 48 minus insulin at entry. Mean and CI come from a linear regression model adjusting for entry insulin, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: Analysis was done in the eligible treated population without insulin use and with data available at all timepoints. The eligible treated population without insulin use includes all participants who received at least one dose of randomized study treatment and who were eligible as per eligibility criteria and were not taking insulin.
Measure: Mean (95% Confidence Interval); unit: μU/ml
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 32 | 40 | 41
μU/ml | 5.20 [-3.29 to 13.70] | 6.02 [-1.57 to 13.62] | -2.86 [-10.4 to 4.66]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting insulin from entry to week 48; Test type: Superiority; p = 0.16, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 8.07, 97.5% CI 2-sided [-4.93 to 21.06] — Mean difference and CI come from a linear regression model adjusting for entry fasting insulin, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.10, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 8.89, 97.5% CI 2-sided [-3.37 to 21.15] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Mean Change (Absolute) in Fasting Insulin From Entry to Week 24
Description: The absolute change is defined as insulin at week 24 minus insulin at entry. Mean and CI come from a linear regression model adjusting for entry insulin, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: μU/ml
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 37 | 42 | 43
μU/ml | 5.86 [-0.96 to 12.68] | 1.95 [-4.47 to 8.37] | 1.57 [-4.78 to 7.93]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in fasting insulin from entry to week 24; Test type: Superiority; p = 0.37, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.28, 97.5% CI 2-sided [-6.42 to 14.99] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.94, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.37, 97.5% CI 2-sided [-10.0 to 10.77] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Mean Change (Absolute) in Insulin Resistance (HOMA-IR) From Entry to Week 48
Description: The absolute change is defined as HOMA-IR at week 48 minus HOMA-IR at entry. HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is a method used to estimate how well the body responds to insulin and is calculated with the following formula: (Fasting insulin, μU/ml)*(Fasting glucose, mg/dL) / 405 Mean and CI come from a linear regression model adjusting for entry HOMA-IR, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: μU/ml
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 32 | 38 | 40
μU/ml | 1.77 [-1.38 to 4.93] | 1.21 [-1.69 to 4.11] | -1.00 [-3.83 to 1.83]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in HOMA-IR from entry to week 48; Test type: Superiority; p = 0.20, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.77, 97.5% CI 2-sided [-2.08 to 7.63] — Mean difference and CI come from a linear regression model adjusting for entry HOMA-IR, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in HOMA-IR from entry to week 48; Test type: Superiority; p = 0.28, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.21, 97.5% CI 2-sided [-2.44 to 6.87] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Mean Change (Absolute) in Insulin Resistance (HOMA-IR) From Entry to Week 24
Description: The absolute change is defined as HOMA-IR at week 24 minus HOMA-IR at entry. HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is a method used to estimate how well the body responds to insulin and is calculated with the following formula: (Fasting insulin, μU/ml)*(Fasting glucose, mg/dL) / 405 Mean and CI come from a linear regression model adjusting for entry HOMA-IR, sex, and race (Black and not Black).
Time Frame: Entry to week 24
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: μU/ml
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 41 | 41
μU/ml | 1.87 [-0.35 to 4.08] | -0.49 [-2.55 to 1.57] | 0.08 [-1.97 to 2.13]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in HOMA-IR from entry to week 24; Test type: Superiority; p = 0.24, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.79, 97.5% CI 2-sided [-1.68 to 5.25] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in absolute change in HOMA-IR from entry to week 24; Test type: Superiority; p = 0.70, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.57, 97.5% CI 2-sided [-3.91 to 2.78] — [estimate comment as in outcome 15, analysis 1]

17. Secondary Outcome: Number of Participants With Confirmed Plasma HIV-1 RNA >200 Copies/mL
Description: Number of participants with confirmed plasma HIV-1 RNA >200 copies/mL, defined as two consecutive results above 200 copies, with the drawing of the second specimen within 2 weeks of site receipt of the first result, and the first result being from a specimen drawn after treatment initiation.
Time Frame: Entry through week 48
Population: Analysis was done in the treated population. This includes all participants who received at least one dose of their randomized study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 47 | 49 | 49
Participants | 0 | 0 | 0

18. Secondary Outcome: Proportion of Participants With Grade ≥3 AEs From Entry to Week 48
Description: Proportion of participants with Grade ≥3 AEs Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Adverse events are graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
Time Frame: Entry to week 48
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 47 | 49 | 49
proportion of participants | 0.23 [0.12 to 0.38] | 0.20 [0.10 to 0.34] | 0.31 [0.18 to 0.45]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in occurrence of Grade ≥3 AEs from entry to week 48; Test type: Superiority; p = 0.43, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in occurrence of Grade ≥3 AEs from entry to week 48; Test type: Superiority; p = 0.26, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value

19. Secondary Outcome: Proportion of Participants With >10% Reduction in Creatinine Clearance (CrCl) From Entry to Week 48
Description: CrCl was estimated by the 2021 CKD-EPI equation and was measured at entry, week 4, week 12, week 24, and week 48.
  The percentage change is defined as CrCl at an on study visit minus CrCl at entry, then divided by CrCl at entry, then multiplied by 100.
  Participants were categorized as experiencing a >10% reduction in CrCl if they experienced the >10% reduction at any of the study visits (week 4, week 12, week 24, and week 48).
Time Frame: Entry to week 48
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 47 | 49 | 49
proportion of participants | 0.23 [0.12 to 0.38] | 0.31 [0.18 to 0.45] | 0.49 [0.34 to 0.64]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in occurrence of >10% reduction in CrCl from entry to week 48; Test type: Superiority; p = 0.008, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 19, analysis 1]; Test type: Superiority; p = 0.068, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value

20. Secondary Outcome: Proportion of Participants With Premature Discontinuation of Study Treatment
Description: Proportion of participants who permanently discontinued any component of study treatment prior to completion of a week 48 visit following randomization
Time Frame: Entry to week 48
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 47 | 49 | 49
proportion of participants | 0.19 [0.09 to 0.33] | 0.14 [0.06 to 0.27] | 0.10 [0.03 to 0.22]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in occurrence of premature discontinuation of study treatment from entry to week 48; Test type: Superiority; p = 0.20, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.56, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; Fisher's Exact Mid P-Value

21. Secondary Outcome: Mean Change (Percent) in Total Fat (kg) From Entry to Week 48
Description: Total fat was measured by DEXA (dual-energy x-ray absorptiometry) scan. The percentage change is defined as total fat at week 48 minus total fat at entry, then divided by total fat at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry total fat, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 42 | 40
relative change % | 0.60 [-2.62 to 3.82] | -2.92 [-5.86 to 0.03] | -2.83 [-5.83 to 0.16]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in total fat from entry to week 48; Test type: Superiority; p = 0.13, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.43, 97.5% CI 2-sided [-1.62 to 8.47] — Mean difference and CI come from a linear regression model adjusting for entry total fat, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in total fat from entry to week 48; Test type: Superiority; p = 0.97, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 97.5% CI 2-sided [-4.89 to 4.72] — [estimate comment as in outcome 21, analysis 1]

22. Secondary Outcome: Mean Change (Percent) in Lean Mass (kg) From Entry to Week 48
Description: Lean mass was measured by DEXA (dual-energy x-ray absorptiometry) scan. The percentage change is defined as lean mass at week 48 minus lean mass at entry, then divided by lean mass at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry lean mass, sex, and race (Black and not Black).
Time Frame: Day 0 to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 42 | 40
relative change % | -1.79 [-3.38 to -0.20] | -0.86 [-2.29 to 0.58] | -2.10 [-3.57 to -0.63]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in lean mass from entry to week 48; Test type: Superiority; p = 0.78, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.31, 97.5% CI 2-sided [-2.18 to 2.80] — Mean difference and CI come from a linear regression model adjusting for entry lean mass, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in lean mass from entry to week 48; Test type: Superiority; p = 0.23, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.24, 97.5% CI 2-sided [-1.11 to 3.59] — [estimate comment as in outcome 22, analysis 1]

23. Secondary Outcome: Mean Change (Percent) in Trunk Fat (kg) From Entry to Week 48
Description: Trunk fat was measured by DEXA (dual-energy x-ray absorptiometry) scan. The percentage change is defined as trunk fat at week 48 minus trunk fat at entry, then divided by trunk fat at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry trunk fat, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 42 | 40
relative change % | 1.32 [-2.63 to 5.26] | -3.75 [-7.34 to -0.15] | -2.39 [-6.07 to 1.28]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in trunk fat from entry to week 48; Test type: Superiority; p = 0.18, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.71, 97.5% CI 2-sided [-2.48 to 9.90] — Mean difference and CI come from a linear regression model adjusting for entry trunk fat, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in trunk fat from entry to week 48; Test type: Superiority; p = 0.60, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.35, 97.5% CI 2-sided [-7.23 to 4.53] — [estimate comment as in outcome 23, analysis 1]

24. Secondary Outcome: Mean Change (Percent) in Limb Fat (kg) From Entry to Week 48
Description: Limb fat was measured by DEXA (dual-energy x-ray absorptiometry) scan. The percentage change is defined as limb fat at week 48 minus limb fat at entry, then divided by limb fat at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry total fat, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 34 | 42 | 39
relative change % | 0.78 [-2.83 to 4.38] | -1.65 [-4.92 to 1.61] | -3.41 [-6.76 to -0.07]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in limb fat from entry to week 48; Test type: Superiority; p = 0.094, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 4.19, 97.5% CI 2-sided [-1.45 to 9.83]; Mean difference and CI come from a linear regression model adjusting for entry limb fat, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in limb fat from entry to week 48; Test type: Superiority; p = 0.46, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 1.76, 97.5% CI 2-sided [-3.59 to 7.11]; [other analysis details as in outcome 24, analysis 1]

25. Secondary Outcome: Mean Change (Percent) in Appendicular Lean Mass (kg) From Entry to Week 48
Description: Appendicular lean mass was measured by DEXA (dual-energy x-ray absorptiometry) scan.
  The percentage change is defined as appendicular lean mass at week 48 minus appendicular lean mass at entry, then divided by appendicular lean mass at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry appendicular lean mass, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 34 | 42 | 39
relative change % | -0.23 [-3.02 to 2.56] | 0.73 [-1.75 to 3.21] | -2.42 [-5.00 to 0.17]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in appendicular lean mass from entry to week 48; Test type: Superiority; p = 0.26, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.19, 97.5% CI 2-sided [-2.19 to 6.56] — Mean difference and CI come from a linear regression model adjusting for entry appendicular lean mass, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 25, analysis 1]; Test type: Superiority; p = 0.084, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.15, 97.5% CI 2-sided [-0.96 to 7.25] — [estimate comment as in outcome 25, analysis 1]

26. Secondary Outcome: Mean Change (Percent) in Hip Bone Mineral Density (g/cm2) From Entry to Week 48
Description: Hip bone mineral density was measured by DEXA (dual-energy x-ray absorptiometry) scan.
  The percentage change is defined as hip bone mineral density at week 48 minus hip bone mineral density at entry, then divided by hip bone mineral density at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry hip bone mineral density, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 40 | 39
relative change % | 0.60 [-0.25 to 1.46] | -0.81 [-1.61 to -0.01] | -0.17 [-0.98 to 0.63]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in hip bone mineral density from entry to week 48; Test type: Superiority; p = 0.19, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.78, 97.5% CI 2-sided [-0.57 to 2.13] — Mean difference and CI come from a linear regression model adjusting for entry hip bone mineral density, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p = 0.27, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.64, 97.5% CI 2-sided [-1.93 to 0.66] — [estimate comment as in outcome 26, analysis 1]

27. Secondary Outcome: Mean Change (Percent) in Lumbar Spine Bone Mineral Density (g/cm2) From Entry to Week 48
Description: Lumbar spine bone mineral density was measured by DEXA (dual-energy x-ray absorptiometry) scan.
  The percentage change is defined as lumbar spine bone mineral density at week 48 minus lumbar spine bone mineral density at entry, then divided by lumbar spine bone mineral density at entry, then multiplied by 100.
  Mean and CI come from a linear regression model adjusting for entry lumbar spine bone mineral density, sex, and race (Black and not Black).
Time Frame: Entry to week 48
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: relative change %
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of INSTI+TAF/FTC
Number analyzed (Participants) | 35 | 42 | 40
relative change % | 0.88 [-0.44 to 2.20] | 0.43 [-0.78 to 1.64] | 0.38 [-0.86 to 1.61]
Statistical Analysis 1: Comparison: DOR 100 mg + TAF/FTC vs Continuation of INSTI+TAF/FTC; Null hypothesis: There is no difference between the two arms in percent change in lumbar spine bone mineral density from entry to week 48; Test type: Superiority; p = 0.58, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.50, 97.5% CI 2-sided [-1.57 to 2.58] — Mean difference and CI come from a linear regression model adjusting for entry lumbar spine bone mineral density, sex, and race (Black and not Black)
Statistical Analysis 2: Comparison: DOR 100 mg + TDF/FTC vs Continuation of INSTI+TAF/FTC; [analysis description as in outcome 27, analysis 1]; Test type: Superiority; p = 0.95, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.05, 97.5% CI 2-sided [-1.93 to 2.03] — [estimate comment as in outcome 27, analysis 1]

ADVERSE EVENTS:
Time Frame: From entry to study completion at Week 48 or premature study discontinuation.
Description: All AEs were recorded on the eCRFs if any of the following criteria were met.
  * All Grade ≥3 AEs
  * All AEs that led to a change in study treatment/intervention regardless of grade
  * All AEs meeting serious adverse event (SAE) definition or expedited adverse event (EAE) reporting requirement
  The DAIDS AE Grading Table (V2.1) was used. All participants who initiated study treatment are included.
Groups:
- DOR 100 mg + TAF/FTC: By mouth daily with or without food. Participants received Doravirine 100 mg tablet by mouth daily. NRTIs (TAF/FTC) were acquired through standard of care locally.
- DOR 100 mg + TDF/FTC: By mouth daily with or without food. Participants received Doravirine 100 mg tablet by mouth daily. NRTIs (TDF/FTC) were acquired through standard of care locally.
- Continuation of Entry INSTI+TAF/FTC: By mouth daily with or without food. INSTIs and NRTIs (TAF/FTC) were acquired through standard of care locally.
Arm/Group | DOR 100 mg + TAF/FTC | DOR 100 mg + TDF/FTC | Continuation of Entry INSTI+TAF/FTC
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 5/47 | 1/49 | 3/49
Other Adverse Events (participants affected / at risk) | 9/47 | 12/49 | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DOR 100 mg + TAF/FTC (N=47) | DOR 100 mg + TDF/FTC (N=49) | Continuation of Entry INSTI+TAF/FTC (N=49)
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DOR 100 mg + TAF/FTC (N=47) | DOR 100 mg + TDF/FTC (N=49) | Continuation of Entry INSTI+TAF/FTC (N=49)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Creatinine renal clearance decreased (Investigations) | 5 | 4 | 8
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 2
Low density lipoprotein increased (Investigations) | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Dependence (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT04636437/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT04636437/SAP_001.pdf